CLINICAL TRIAL: NCT05116449
Title: Comparison of Changes in the Quality of Life of Patients Operated on Breast Cancer at the Drôme Ardèche Breast Institute According to Access to Supportive Oncological Care
Brief Title: Comparison of Changes in the Quality of Life of Patients Operated on Breast Cancer at the Drôme Ardèche Breast Institute According to Access to Supportive Oncological Care (IDSein)
Acronym: IDSein
Status: Recruiting | Type: Observational
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: European Clinical Trial Experts Network (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-A02397-50
Record Dates: First submitted 2021-11-04; First posted 2021-11-11 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patient seeking supportive care
  Interventions: Behavioral: Quality of life questionnaires
- Patient without any supportive care
  Interventions: Behavioral: Quality of life questionnaires

INTERVENTIONS:
Behavioral: Quality of life questionnaires — Different quality of life questionnaires : FACT-B, EORTC QLQ-C30, QIC, BRIEF COPE, HADS, QSSS-C

SUMMARY:
The aim of this study is to explore the quality of life of cancer patients, in particular women operated on breast cancer, throughout their care journey, taking into account their access to supportive oncological care within and outside the establishment care.

ELIGIBILITY:
Inclusion Criteria:

* Woman with histologically confirmed invasive breast cancer for whom surgery is scheduled
* Age> 18 years old
* Performance status ECOG <2
* Patient speaking and understanding French and able to complete questionnaires
* Patient affiliated or beneficiary of a social security scheme
* Patient having read the information note and not objecting to the use of the data collected

Exclusion Criteria:

* male
* Patient with metastatic breast cancer
* Patient with bilateral breast cancer
* History of cancer of less than 5 years
* Active infection or other serious underlying condition that may prevent the patient from receiving treatment
* History or progressive psychiatric illness
* Person deprived of liberty or under guardianship
* Inability to undergo medical monitoring for geographical, social or psychological reasons Indication of emergency amputation
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision
* Pregnant, breastfeeding or parturient woman
* Patient hospitalized without consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women patient with breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2021-02-22 (Actual); Primary Completion 2025-12-22 (Estimated); Study Completion 2026-01-22 (Estimated)

PRIMARY OUTCOMES:
Quality of life questionnaire : FACT-B | 12 months
  Functional Assessment of Cancer Therapy-breast : 27 items about physical well-being, family well-being, emotional and functional well-being. The quotation is between 0 "not at all" and 4 "verry much". The total score is between 0 and 148.
  The higher the scores, the higher the QoL and the various well-being.
Quality of life questionnaire : EORTC QLQ-C30 | 12 months
  30 items for all patient suffering from cancer. The answer of each question is between 1 "not at all" and 4 "very much"

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Institut du sein Drôme Ardèche, Guilherand-Granges
  - Hôpital Privé de l'Estuaire, Le Havre